CLINICAL TRIAL: NCT05785650
Title: Trigger Points of Supraspinatus Muscle: Osteopaths' Palpation Reproductibility and Ultrasound Translation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Institut des Hautes Etudes Osteopathiques de Nantes (Other)
Responsible Party: Sponsor
Other Study IDs: TRIGGOSTEO-1; 2023-A00637-38 (Other: Agence nationale de sécurité du médicament et produits de santé)
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Shoulder Pain
Keywords: trigger point; osteopathic palpation; ultrasound
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: osteopathic palpation — comparaison of ultrasound caracteristics of areas with ad without TP

SUMMARY:
Trigger points (TP) are described as "hard, palpable nodules located within the taut bands of skeletal muscle" (Bardoni, 2022).

The aim of this study is to evaluate the reproductibility of palpation of TP between osteopaths and to compare this perception to ultrasound measures of echogenicity.

Method:

A sample of 61 patients will be included in the study. An osteopath will determine the eligibility of the study. The supraclavicular area will be mark every 2 cm to establish a grid for all evaluations.

First an osteopath will evaluate with palpation the presence of TP at every box of the grid.

A second osteopath will evaluate the same boxes and will be blinded to the result of the first osteopath.

At each step of palpation, a pain assessment will be carried out at each box. Then, the ultrasound technician will evaluate the echogeneicity of every box and will be blinded to the prior results.

The protocol will be approve by a french ethic committee.

DETAILED DESCRIPTION:
sensitivity and specificity of osteopathic tests will be conducted in comparaison to echograph results (a binary outcomes assessing the presence of an hypoechogenicity).

The reproductibility of osteopaths' tests will be be calculated using Cohen's kappa weighted by the distance between the TPs found.

Finally, the pain reported by patients on areas with a TP defined by the osteopath, and the pain reported by patients on areas without a TP defined by the osteopath will be compared using a student test.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 to 50 years old),
* affiliation to a social security scheme or beneficiary of such a scheme

Exclusion Criteria:

* pregnant and breastfeeding women,
* adults under guardianship and protected patients.
* History of integumentary or muscular involvement in the area of interest
* Allergic reaction
* wish to stop the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: There will be 61 healthy adults The population studied will be heterogeneous with or without shoulder pain Recruitment will be based on students or patients of IdHEO Nantes osteopathy clinic on a voluntary basis.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Estimated)
Dates: Start 2023-08-30 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
sensitivity and specificity of osteopathic tests | at day 1
  to compare osteopath TP detection to ultrasound echogenicity

SECONDARY OUTCOMES:
Inter examiner reproductibility of TP detection | at day 1
  using Cohen's kappa weighted by the distance between the TPs found. Quadratic weighting will be used.
camparison of pain reported by patient with TP detection by osteopath | at day 1
  using a student test between pain means in areas with and without TP

IPD SHARING:
Plan to Share IPD: Yes
on demand to m. salmon
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code